CLINICAL TRIAL: NCT05863715
Title: Working Memory Quality of Attentional Templates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-05-03; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: attention; visual search; working memory

STUDY DESIGN:
Intervention Model Description: All participants receive each level of visual cue type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-subjects Cue Type (Experimental): Participants receive a target color cue (positive), a distractor color cue (negative), or a neutral non-informative cue prior to visual search.
  Interventions: Behavioral: Visual Search Cue Type

INTERVENTIONS:
Behavioral: Visual Search Cue Type — Participants receive a target color cue (positive), a distractor color cue (negative), or a neutral non-informative cue prior to visual search.

SUMMARY:
In this line of research, the researchers are examining a basic science question regarding the working memory representations underlying visual search using a positive template (looking for a target) or a negative template (avoiding a distractor).

DETAILED DESCRIPTION:
When finding a search target, receiving a target cue or distractor cue can increase search efficiency. Critically, in order to use these cues to help search performance, they must be maintained in working memory. The researchers are examining whether the working memory representations are of similar quality for a target cue (positive template) or distractor cue (negative template).

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Button Press Reaction Time | Day 1 (single day of testing)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | Day 1 (single day of testing)
  Accuracy of responses to target item-measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button
Working Memory Report Quality | Day 1 (single day of testing)
  Accuracy of computer clicks on a set of colors to indicate memory of cue presented

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.